CLINICAL TRIAL: NCT01482598
Title: COR HF - Clinical Benefits in Optimized Remote HF Patient Management
Brief Title: Clinical Benefits in Optimized Remote HF Patient Management
Acronym: COR-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR-11-017-IT-HF
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Congestive Heart Failure Treated
Keywords: Heart Failure; Cardiac Resynchronization Therapy; Remote Care; Disease Management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimal Remote Care (Active Comparator): Patient follow up is performed through remote care, remote alerts on CRT-D device data are transmitted daily to the hospital, remote follow up is scheduled every 6 months, hospital in clinic follow up is scheduled at 12 months after implant.
  Interventions: Device: Remote Care Follow up
- Optimal Standard Care (No Intervention): Patient standard in clinic visits are performed every 6 months.

INTERVENTIONS:
Device: Remote Care Follow up — Patient device is checked daily through remote transmitter (Merlin@Home) and every 6 month a complete transmission with all device data is performed
  Other Names: Home monitoring, Remote monitoring, Merlin.net
  Arms: Optimal Remote Care

SUMMARY:
The Study Purpose is to demonstrate the superiority of optimized remote patient management compared to optimized standard care in the management and prognosis of heart failure, in the prevention of recurrent atrial tachycardia or atrial fibrillation episodes and in the reduction of inappropriate shock therapies. The remote care allows early intervention in terms of drug therapy adjustment and cardiac resynchronization therapy (CRT-D) device reprogramming.

DETAILED DESCRIPTION:
The outcome measure of the study is a combined endpoint of:

* Proportion of patients with HF hospitalization or emergency unit admission with intravenous diuretics, Atrial Tachycardia/Atrial Fibrillation (AT/AF) episodes or cardiovascular/cerebrovascular episodes requiring hospitalization at 12 months
* Proportion of patients with inappropriate Implantable Cardioverter-Defibrillator (ICD) therapies delivered at 12 months comparing optimized remote patient management to optimized standard patient management

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients already implanted with CRT-D devices (from 4 to 8 weeks), according to current guidelines1
* 1 hospitalization or access to emergency unit due to heart failure (including treatment with diuretic and/or cardioactive intravenous therapy) within the last 12 months
* Left Bundle Branch Block (LBBB)
* Patients must be able to provide written informed consent
* Patients are mentally capable to participate in the Investigation (based on physician's discretion)

Exclusion Criteria:

* Patients already implanted with CRT or CRT-D device to be replaced
* Patients in long-standing persistent or permanent AT/AF
* Patients in dialysis treatment at the time of enrollment
* Patients in parenteral inotropic therapy at the time of enrollment
* Patients with epicardial Left Ventricular (LV) lead
* Patients with mechanical valvular prosthesis
* Patients with life expectancy < 12 months
* Patients actively considered for cardiac transplant
* Patients < 18 years old
* Pregnant women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2011-10; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Padeletti, Prof., Study Chair — Azienda Ospedaliero-Universitaria Careggi; Maria Grazia Bongiorni, MD, Principal Investigator — Ospedale S.Chiara-Cisanello, Pisa; Gerardo Ansalone, MD, Principal Investigator — Ospedale Vannini, Roma; Gianluca Botto, MD, Principal Investigator — Ospedale S. Anna, Como; Antonio Curnis, MD, Principal Investigator — Spedali Civili, Brescia; Stefano Favale, Prof., Principal Investigator — Policlinico Consorziale, Bari; Edoardo Gronda, MD, Principal Investigator — Multimedica IRCCS, Milano; Roberto Verlato, MD, Principal Investigator — Ospedale Pietro Cosma, Camposampiero (PD); Alessandro Proclemer, MD, Principal Investigator — Ospedale S.M. della Misericordia, Udine; Luca Santini, MD, Principal Investigator — University of Rome Tor Vergata; Alessandro Capucci, Prof., Principal Investigator — Azienda Ospedaliero, Universitaria Ospedali Riuniti; Francesco Solimene, MD, Principal Investigator — Casa di Cura "Montevergine", Mercogliano (AV)
Locations (18):
- Italy (18):
  - Casa di Cura "Montevergine", Mercogliano, Avellino
  - Ospedale Pietro Cosma, Camposampiero, Padova
  - Osp. S.Raffaele Giglio, Cefalù, Palermo
  - Presidio Ospedaliero Riunito di Ciriè, Cirié, Torino
  - Presidio Ospedaliero di Conegliano, Conegliano, Treviso
  - Casa di Cura Pederzoli, Peschiera del Garda, Verona
  - Azienda Ospedaliero Universitaria "Ospedali Riuniti", Ancona
  - Policlinico Consorziale, Bari
  - Spedali Civili, Brescia
  - Ospedale Ferrarotto Vittorio Emanuele, Catania
  - Ospedale S. Anna, Como
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliera dei Colli - Ospedale Monaldi, Napoli
  - Ospedale Guglielmo da Saliceto, Piacenza
  - Ospedale S. Chiara - Cisanello, Pisa
  - Ospedale Vannini, Roma
  - Policlinico Tor Vergata, Roma
  - Ospedale di Belcolle, Viterbo

REFERENCES:
- [Background] Santini M, Ricci RP, Lunati M, Landolina M, Perego GB, Marzegalli M, Schirru M, Belvito C, Brambilla R, Guenzati G, Gilardi S, Valsecchi S. Remote monitoring of patients with biventricular defibrillators through the CareLink system improves clinical management of arrhythmias and heart failure episodes. J Interv Card Electrophysiol. 2009 Jan;24(1):53-61. doi: 10.1007/s10840-008-9321-3. Epub 2008 Oct 31. PMID 18975066
- [Background] Marzegalli M, Lunati M, Landolina M, Perego GB, Ricci RP, Guenzati G, Schirru M, Belvito C, Brambilla R, Masella C, Di Stasi F, Valsecchi S, Santini M. Remote monitoring of CRT-ICD: the multicenter Italian CareLink evaluation--ease of use, acceptance, and organizational implications. Pacing Clin Electrophysiol. 2008 Oct;31(10):1259-64. doi: 10.1111/j.1540-8159.2008.01175.x. PMID 18811805
- [Background] Abraham WT, Compton S, Haas G, Foreman B, Canby RC, Fishel R, McRae S, Toledo GB, Sarkar S, Hettrick DA; FAST Study Investigators. Intrathoracic impedance vs daily weight monitoring for predicting worsening heart failure events: results of the Fluid Accumulation Status Trial (FAST). Congest Heart Fail. 2011 Mar-Apr;17(2):51-5. doi: 10.1111/j.1751-7133.2011.00220.x. Epub 2011 Mar 21. PMID 21449992
- [Background] Abraham WT, Gras D, Yu CM, Guzzo L, Gupta MS; FREEDOM Steering Committee. Rationale and design of a randomized clinical trial to assess the safety and efficacy of frequent optimization of cardiac resynchronization therapy: the Frequent Optimization Study Using the QuickOpt Method (FREEDOM) trial. Am Heart J. 2010 Jun;159(6):944-948.e1. doi: 10.1016/j.ahj.2010.02.034. PMID 20569704
- [Background] Chaudhry SI, Mattera JA, Curtis JP, Spertus JA, Herrin J, Lin Z, Phillips CO, Hodshon BV, Cooper LS, Krumholz HM. Telemonitoring in patients with heart failure. N Engl J Med. 2010 Dec 9;363(24):2301-9. doi: 10.1056/NEJMoa1010029. Epub 2010 Nov 16. PMID 21080835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 subjects not randomized. 139 Subjects randomized in 2 arms
Period: Overall Study
Arm/Group | Optimal Remote Care | Optimal Standard Care
Started (1st subject was enrolled on 19th October 2011) | 66 | 73
Completed (last subject was enrolled on 9th June 2014) | 50 | 51
Not Completed | 16 | 22
Not completed — Death | 7 | 10
Not completed — Physician Decision | 0 | 3
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Optimal Remote Care: Patient follow up is performed through remote care, remote alerts on Cardiac Resynchronization Therapy - Defibrillator (CRT-D) device data are transmitted daily to the hospital, remote follow up is scheduled every 6 months, hospital in clinic follow up is scheduled at 12 months after implant.
  Remote Care Follow up: Patient device is checked daily through remote transmitter (Merlin@Home) and every 6 month a complete transmission with all device data is performed
- Total: Total of all reporting groups
Arm/Group | Optimal Remote Care | Optimal Standard Care | Total
Number analyzed (Participants) | 66 | 73 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (11.3) | 71.9 (10.6) | 71.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 49 | 53 | 102
Weight (kg) [Mean (Standard Deviation); unit: Kg] — Population: Weight in Remote Care Arm was available only for 65 subjects instead of 66.
  Kg
    number analyzed (Participants) | 65 | 73 | 138
    (all) | 76.1 (15.5) | 74.4 (14.3) | 75.2 (14.8)
Height (cm) [Mean (Standard Deviation); unit: cm] — Population: info not available for the entire population
  cm
    number analyzed (Participants) | 64 | 71 | 135
    (all) | 169.0 (7.8) | 168.5 (8.0) | 168.7 (7.9)
NYHA Class [Number; unit: participants] — New York Heart Association (NYHA) functional classification for heart failure. It places patients in four categories based on the limitation during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina pain.
  Class I: Cardiac disease without limitation of physical activity. Class II: Cardiac disease with slight limitation of physical activity. Class III: Cardiac disease with marked limitation of physical activity. Class IV: Cardiac disease with inability to carry on any physical activity without discomfort.
  participants
    NYHA Class I | 5 | 4 | 9
    NYHA Class II | 24 | 27 | 51
    NYHA Class III | 35 | 41 | 76
    NYHA Class IV | 2 | 1 | 3
Widest Intrinsic Complex (QRS) duration (msec) [Mean (Standard Deviation); unit: msec] — data not available for the entire population Population: Data not available for the entire study population
  msec
    number analyzed (Participants) | 62 | 72 | 134
    (all) | 155.9 (23.5) | 152.5 (22.9) | 154.0 (23.2)
Current Medication [Count of Participants; unit: Participants]
  Beta Blockers | 53 | 60 | 113
  Angiotensin-Converting Enzyme (ACE) Inhibitors | 40 | 49 | 89
  Diuretics | 63 | 66 | 129
  Aldosterone Antagonist | 23 | 24 | 47
  Angiotensin Receptor Blockers (ARBs) | 13 | 16 | 29
  Amiodarone | 12 | 15 | 27
  Other Antiarrhythmics | 1 | 3 | 4
  Statins | 35 | 32 | 67
  Cardiac Glycosides | 6 | 3 | 9
  Other | 57 | 64 | 121
Etiology of cardiovascular disease (Ischemic/Non Ischemic) [Count of Participants; unit: Participants]
  Ischemic | 31 | 27 | 58
  Non Ischemic | 35 | 44 | 79
Comorbidities [Count of Participants; unit: Participants]
  None | 2 | 7 | 9
  Paroxysmal AT/AF | 6 | 10 | 16
  Hypertension | 38 | 38 | 76
  Hypercholesterolemia | 26 | 16 | 42
  Diabetes Mellitus | 14 | 19 | 33
  Chronic Obstructive Pulmonary Disease | 8 | 13 | 21
  Chronic Renal Insufficiency | 8 | 9 | 17
  Dysthyroidism | 5 | 5 | 10
  Smoking | 32 | 29 | 61
  Other | 14 | 24 | 38
Implant Information [Count of Participants; unit: Participants]
  Implantation Indication (Primary Prevention) | 60 | 65 | 125
  Implantation Indication (Secondary Prevention) | 6 | 8 | 14
  Pulse Generator (CRT-D) Position (Left) | 64 | 72 | 136
  Pulse Generator (CRT-D) Position (Right) | 2 | 1 | 3
  RA Lead Position (Atrial Appendage) | 65 | 69 | 134
  RA Lead Position (Atrial Septum) | 0 | 3 | 3
  RA Lead Position (Atrial Freewall) | 1 | 0 | 1
  RA Lead Position (Other) | 0 | 1 | 1
  RV Lead Position (RV Apex) | 38 | 41 | 79
  RV Lead Position (RV Septum) | 25 | 31 | 56
  RV Lead Position (RV Outflow) | 2 | 1 | 3
  RV Lead Position (Other) | 1 | 0 | 1
  Left Ventricle (LV) Lead Tip Position (Basal Anterior) | 2 | 0 | 2
  LV Lead Tip Position (Basal Lateral) | 7 | 11 | 18
  LV Lead Tip Position (Basal Posterior) | 7 | 2 | 9
  LV Lead Tip Position (Basal Inferior) | 0 | 0 | 0
  LV Lead Tip Position (Basal Post. Septum) | 0 | 0 | 0
  LV Lead Tip Position (Basal Ant. Septum) | 0 | 0 | 0
  LV Lead Tip Position (Medium Anterior) | 1 | 0 | 1
  LV Lead Tip Position (Medium Lateral) | 35 | 46 | 81
  LV Lead Tip Position (Medium Posterior) | 13 | 14 | 27
  LV Lead Tip Position (Medium Inferior) | 0 | 0 | 0
  LV Lead Tip Position (Medium Post Septum) | 1 | 0 | 1
  LV Lead Tip Position (Medium Ant Septum) | 0 | 0 | 0
  Final Programmed LV Configuration (Distal 1 - Mid 2) | 26 | 29 | 55
  Final Programmed LV Configuration (Distal 1 - Prox 4) | 2 | 5 | 7
  Final Programmed LV Configuration (Distal 1 - RV Coil) | 7 | 11 | 18
  Final Programmed LV Configuration (Mid 2 - Prox 4) | 3 | 3 | 6
  Final Programmed LV Configuration (Mid 2 - RV Coil) | 6 | 9 | 15
  Final Programmed LV Configuration (Mid 3 - Mid 2) | 6 | 3 | 9
  Final Programmed LV Configuration (Mid 3 - Prox 4) | 7 | 3 | 10
  Final Programmed LV Configuration (Mid 3 - RV Coil)) | 5 | 5 | 10
  Final Programmed LV Configuration (Prox 4 - Mid 2) | 1 | 1 | 2
  Final Programmed LV Configuration (Prox 4 - RV Coil) | 3 | 4 | 7
Implant Information (Electrical Measures) [Mean (Standard Deviation); unit: units on a scale] — Population: Measure Description: data not available for the entire population
  units on a scale
    Capture Threshold (V) at 0.5 ms: number analyzed (Participants) | 66 | 72 | 138
    Capture Threshold (V) at 0.5 ms | 14 (0.8) | 1.4 (1.1) | 1.4 (1.0)
    Phrenic Nerve Stimulation Threshold (V) at 0.5 ms: number analyzed (Participants) | 4 | 5 | 9
    Phrenic Nerve Stimulation Threshold (V) at 0.5 ms | 4.6 (1.4) | 4.9 (1.6) | 4.8 (1.4)
Implant Information (Electrical Measures) [Mean (Standard Deviation); unit: Impedance (Ω)] — Measure Analysis Population Description: data not available for the entire population
  Impedance (Ω) | 773.3 (259.3) | 757.1 (237.2) | 764.8 (247.1)
Implant Information (AV/PV & V-V Delay Optimization method) [Count of Participants; unit: Participants] — Atrioventricular (AV/PV) and interventricular (VV) delay optimization in pacing devices can be performed using different methods.
  Echo: standard AV/PV and/or VV delay optimization guided by Doppler echocardiogram measurements of the maximum aortic velocity time integral (aortic VTI).
  Echo (Specify parameters): AV/PV and/or VV delay optimization guided by Doppler according to specific parameters.
  Automated Optimization (QuickOpt™): proprietary algorithm for AV/PV and VV delay optimization based on intracardiac electrogram (IEGM) measurement.
  Default Parameters: Standard device parameters.
  Participants
    Echo | 0 | 4 | 4
    Echo (Specify parameters) | 0 | 2 | 2
    QuickOpt | 39 | 32 | 71
    Default Parameters | 15 | 23 | 38
    Other | 12 | 12 | 24
Implant Information (Device Programming) [Count of Participants; unit: Participants]
  Pacing Mode (DDD) | 66 | 73 | 139
  Sensor (On) | 6 | 6 | 12
  Sensor (Off) | 60 | 67 | 127
  AF Suppression (On) | 0 | 0 | 0
  AF Suppression (Off) | 66 | 73 | 139
Implant Information (Base Rate) [Mean (Standard Deviation); unit: bpm] — Measure Analysis Population Description: data not available for the entire population
  bpm | 52.5 (7.4) | 52.7 (7.8) | 52.6 (7.6)
Implant Information (Intervals Programming) [Mean (Standard Deviation); unit: units on a scale] — Population: data not available for the entire population
  units on a scale
    AV Delay (msec) | 147.4 (24.3) | 146.2 (18.3) | 146.8 (21.3)
    PV Delay (msec) | 112.1 (14.4) | 111.8 (13.3) | 111.9 (13.8)
    VV Delay (msec): number analyzed (Participants) | 36 | 47 | 83
    VV Delay (msec) | 34.4 (15.2) | 33.7 (15.9) | 34.0 (15.5)
Implant Information (VV Delay and Final LV Pacing Vector Programming) [Count of Participants; unit: Participants] — The VV Delay is the interval between right ventricular (RV) and left ventricular (LV)activation; Simultaneous (VV Delay = 0), LV First (left pre-activation) o RV First (right pre-activation) are programmable configurations. In addition the LV Pacing Vector is programmable in 10 different configurations to optimize the LV contraction and the resynchronization of the two ventricles.
  Participants
    VV Delay (Simultaneous) | 30 | 26 | 56
    VV Delay (LV First) | 34 | 46 | 80
    VV Delay (RV First) | 2 | 1 | 3
    Final LV Pacing Vector (Distal 1 - Mid 2) | 26 | 30 | 56
    Final LV Pacing Vector (Distal 1 - Prox 4) | 2 | 5 | 7
    Final LV Pacing Vector (Distal 1 - RV Coil) | 7 | 11 | 18
    Final LV Pacing Vector (Mid 2 - Prox 4) | 3 | 3 | 6
    Final LV Pacing Vector (Mid 2 - RV Coil) | 6 | 10 | 16
    Final LV Pacing Vector (Mid 3 - Mid 2) | 6 | 3 | 9
    Final LV Pacing Vector (Mid 3 - Prox 4) | 7 | 3 | 10
    Final LV Pacing Vector (Mid 3 - RV Coil) | 5 | 4 | 9
    Final LV Pacing Vector (Prox 4 - Mid 2) | 1 | 0 | 1
    Final LV Pacing Vector (Prox 4 - RV Coil) | 3 | 4 | 7
Implant Information (Patient Notifier and Merlin.net Programming) [Count of Participants; unit: Participants] — Data not available for the entire study population Population: data not available for the entire population
  Participants
    Patient Notifier programmed as Protocol: Yes | 63 | 67 | 130
    Patient Notifier programmed as Protocol: No | 3 | 6 | 9
    Merlin.Net patient profile programmed as Protocol: Yes | 65 | 5 | 70
    Merlin.Net patient profile programmed as Protocol: No | 1 | 68 | 69
    Direct Alerts programmed as Protocol: number analyzed (Participants) | 65 | 5 | 70
    Direct Alerts programmed as Protocol: Yes | 65 | 5 | 70
    Direct Alerts programmed as Protocol: No | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Combined Endpoint on Patient Clinical Outcome
Description: Combined Endpoint:
  * proportion of patients with HF hospitalization or emergency unit admission with intravenous diuretics, Atrial Tachycardia/Atrial Fibrillation (AT/AF) episodes or cardiovascular/cerebrovascular episodes requiring hospitalization at 12 months
  * proportion of patients with inappropriate Implantable Cardiac Defibrillator (ICD) therapies delivered at 12 months
Time Frame: 12 months follow up
Population: The study enrolled less than one third of expected patients as per sample size (144 out of 438). The pool of data collected during the follow up phase were spare and incomplete for the major part of patients enrolled. In addition an high number of deviations were collected during the study due to incomplete data collection. For the aforementioned reasons, the analysis for primary and secondary endpoints hasn't been performed.
Groups:
- Remote Care: Patients perform a 6 and 18 (optional) months Remote Follow Up and 12 and 24 months in clinic visits
Arm/Group | Optimal Standard Care | Remote Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Optimal Standard Care | Remote Care
All-Cause Mortality (participants affected / at risk) | 10/73 | 8/66
Serious Adverse Events (participants affected / at risk) | 37/73 | 28/66
Other Adverse Events (participants affected / at risk) | 13/73 | 21/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimal Standard Care (N=73) | Remote Care (N=66)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 1 (1)
Heart Failure (Cardiac disorders) | 10 (13) | 7 (8)
Pulmonary Edema (Cardiac disorders) | 1 (1) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac Death (General disorders) | 1 (1) | 0 (0)
Infected Skin Ulcer (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Implant Site Infection (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Respiratory Failure (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Carotid Artery Thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Colonic Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Coxarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Non ST segment elevation acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Hemodynamic Instability (General disorders) | 0 (0) | 1 (1)
Sudden Death, Cause Unknown (Cardiac disorders) | 1 (1) | 0 (0)
Unknown Cause of Death (General disorders) | 1 (1) | 0 (0)
Pocket Formation of Decubitus (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Medical Device Replacement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Renal Venous Congestion (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteomyelitis of the foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer Metastatic (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic Valve Replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Foot Amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin Graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiogenic Shock (Vascular disorders) | 0 (0) | 1 (1)
Lead Dislodgement (Product Issues) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimal Standard Care (N=73) | Remote Care (N=66)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnea (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary Congestion (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary Edema (Cardiac disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest Crushing (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Angiogram (Investigations) | 0 (0) | 1 (1)
Sinus Rhythm (Investigations) | 1 (1) | 0 (0)
Device Capturing Issue (Product Issues) | 1 (1) | 4 (4)
Device Electrical Impedance Issue (Product Issues) | 1 (1) | 1 (1)
Device Inappropriate shock delivery (Product Issues) | 2 (2) | 4 (4)
Device Malfunction (Product Issues) | 1 (1) | 2 (2)
Device Telemetry Issue (Product Issues) | 0 (0) | 2 (2)
Lead Dislodgement (Product Issues) | 1 (1) | 0 (0)
Mobile Medical Application Issue (Product Issues) | 0 (0) | 1 (1)
Oversensing (Product Issues) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No